CLINICAL TRIAL: NCT04158427
Title: Intestinal Microbiota and Chronic Fatigue Syndrome. Effect of Fecal Transplant on Health Related Quality of Life of the Patients With Chronic Fatigue Syndrome
Brief Title: Intestinal Microbiota and Chronic Fatigue Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Tapani Salonen, Principal Investigator, MD, PhD, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R18006
Record Dates: First submitted 2019-08-08; First posted 2019-11-08 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Fatigue Syndrome, Chronic; Microbial Colonization
Keywords: fatigue; microbiome
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Communicable Diseases; Fatigue | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Double-blinded study, treatment group and placebo-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded products, investigators and patients are blinded. Fecal transplant is either from a healthy donor or patient's own feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal transplant (Experimental): A single dose fecal transplant is given (via colonoscopy) from a healthy donor
  Interventions: Procedure: Faecal transplantation
- Placebo (Placebo Comparator): A single dose patient's own feces is given (via colonoscopy)
  Interventions: Procedure: Placebo faecal transplantation

INTERVENTIONS:
Procedure: Faecal transplantation — Faecal transplantation from a healthy donor via colonoscopy
  Arms: Fecal transplant
Procedure: Placebo faecal transplantation — Placebo faecal transplantation containing patient's own feces via colonoscopy
  Arms: Placebo

SUMMARY:
Gut microbiota of 1) patients with chronic fatigue syndrome and 2) their healthy family members are analyzed.

Up to 40 patients with chronic fatigue syndrome are randomized to receive either 1) a faecal transplant from a healthty donor or 2) their own feces via colonoscopy. Patient's health related quality and ability to work are assessed (baseline, 1 and 6 months after the procedure)

DETAILED DESCRIPTION:
Patients with chronic fatigue syndrome (CFS) and their healthy family members (living together in the same house) are recruited in the study. CFS has been diagnosed in Tampere University Hospital and the diagnosis is based on thorough clinical assessment fulfilling the Institute of Medicine 2015 criteria. Patients microbiota is analyzed (microbiological analysis, mediators of inflammation) and results are compared with their family members.

Via colonoscopy, up to 40 patients with CFS are randomized to receive either a faecal transplant from a healthy donor (treatment group) or his/her own feces (placebo group). Products are blinded, investigators and patients are blinded. Patients' health related quality of life and ability to work or study are assessed (baseline, 1 and 6 months after the procedure).

ELIGIBILITY:
Inclusion Criteria:

-Chronic Fatigue Syndrome

Exclusion Criteria:

* Other conditions causing chronic fatigue
* Diseases affecting the intestinal system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Health related quality of life assessed by EQ-5D-5L questionnaire | Change from Baseline EQ-5D-5L scores at 6 months after the procedure
  Health related quality of life, Euro-QoL 5 Dimension (EQ-5D-5L scores) (5 levels of perceived problems, scale from 1 (no problems/the best) to 5 (extreme problems/unable to)
Health related quality of life assessed by 15D questionnaire | Change from Baseline 15D scores at 6 months after the procedure
  Health related quality of life, 15D scores (15 separate dimensions, scale from 1 to 5; 1=the highest/best level), 5=the lowest/worst level)
Health related quality of life assessed by Modified Fatigue Impact Scale | Change from Baseline Modified Fatigue Impact Scale scores at 6 months after the procedure
  Health related quality of life, Modified Fatigue Impact Scale scores (Total Score, range 0 to 84; Physical subscale, range 0 to 36; Cognitive Subscale, range 0 to 40; Psychosocial Subscale, range from 0 to 8 (0 = no fatigue, highest points = extreme fatigue)
Ability to work or study | Change from Baseline at 6 months after the procedure
  Whether ability to work or study has been restored (value is 1) or not (value is 0)
Visual Analog Fatigue Scale | Change from Baseline Visual Analog Fatigue Scale point at 6 months after the procedure
  A 100 mm horizontal line with written descriptions at each end (0 = no fatigue; 100 = extreme fatigue)

SECONDARY OUTCOMES:
Health related quality of life assessed by EQ-5D-5L questionnaire | Change from Baseline EQ-5D-5L scores at 1 months after the procedure
  Health related quality of life, Euro-QoL 5 Dimension (EQ-5D-5L scores) (5 levels of perceived problems, scale from 1 (no problems/the best) to 5 (extreme problems/unable to)
Health related quality of life assessed by 15D questionnaire | Change from Baseline 15D at 1 months after the procedure
  Health related quality of life, 15D scores (15 separate dimensions, scale from 1 to 5; 1=the highest/best level), 5=the lowest/worst level)
Health related quality of life assessed by Modified Fatigue Impact Scale | Change from Baseline Modified Fatigue Impact Scale scores at 1 months after the procedure
  Health related quality of life, Modified Fatigue Impact Scale scores (Total Score, range 0 to 84; Physical subscale, range 0 to 36; Cognitive Subscale, range 0 to 40; Psychosocial Subscale, range from 0 to 8 (0 = no fatigue, highest points = extreme fatigue)
Ability to work or study | Change from Baseline at 1 months after the procedure
  Whether ability to work or study has been restored (value is 1) or not (value is 0)
Visual Analog Fatigue Scale | Change from Baseline Visual Analog Fatigue Scale point at 1 months after the procedure
  A 100 mm horizontal line with written descriptions at each end (0 = no fatigue; 100 = extreme fatigue)

CONTACTS AND LOCATIONS:
Overall Officials: Tapani Salonen, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salonen T, Jokinen E, Satokari R, Lahtinen P. Randomized, double-blinded, placebo-controlled pilot study: efficacy of faecal microbiota transplantation on chronic fatigue syndrome. J Transl Med. 2023 Jul 29;21(1):513. doi: 10.1186/s12967-023-04227-y. PMID 37516837